CLINICAL TRIAL: NCT03279224
Title: A Randomized Controlled Trial of the Safety and Efficacy of Fecal Microbiota Transplantation in a Population With Bipolar Disorder
Brief Title: Safety and Efficacy of Fecal Microbiota Transplantation in a Population With Bipolar Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Valerie Taylor (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Valerie Taylor, Psychiatrist-in-Chief, Women's College Hospital
Organization: Women's College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAN-FMT-WCH-2016
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Bipolar Depression
Keywords: Bipolar, Depression, FMT, Microbiome
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Adults with BD depression being treated with an approved medication will be assigned to either allogenic FMT (from a healthy, screened individual with no personal or family history of an Axis 1 disorder) or autologous FMT (re-infusion of own feces)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the patient and the study team (clinical team, study coordinator, data analyst) will be blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic FMT (Active Comparator): Participants Randomized to this arm will receive FMT (Fecal Microbiota Transplantation) from a healthy, screened individual with no personal or family history of an Axis 1 disorder.
  Interventions: Biological: Allogenic FMT
- Autologous FMT (Placebo Comparator): Participants Randomized to this arm will receive FMT (Fecal Microbiota Transplantation) by re-infusion of their own feces donated earlier in the study.
  Interventions: Biological: Autologous FMT

INTERVENTIONS:
Biological: Allogenic FMT — Fifty (50) g of screened donor feces will be weighed and homogenized with 30 mL of sterile 0.9 N NaCl + 10% glycerol using a sterile 330 micron micro-filter-separated double-compartment polyethylene bag in the Stomacher® Paddle Blender.
  2.The volume of fecal filtrate corresponding to fifty (50) g of donor stools will be transferred into a 50 mL Falcon tube with screw top and frozen at -80oC.
  3. For colonoscopy administration, three (3) Falcon tubes of thawed FMT concentrated will be diluted to a total volume of 300 mL with 0.9N NaCl and will be transported to the endoscopy suite. In the endoscopy suite, the FMT product will be packaged into 6 x 50 ml syringes for patient delivery by colonoscopy.
  Arms: Allogenic FMT
Biological: Autologous FMT — 1. Fifty (50) g of the participant's feces will be weighed and homogenized with 30 mL of sterile 0.9 N NaCl + 10% glycerol using a sterile 330 micron micro-filter-separated double-compartment polyethylene bag in the Stomacher® Paddle Blender.
  3.The volume of fecal filtrate corresponding to fifty (50) g of participant's stools will be transferred into a 50 mL Falcon tube with screw top and frozen at -80oC.
  3. For colonoscopy administration, three (3) Falcon tubes of thawed FMT concentrated will be diluted to a total volume of 300 mL with 0.9N NaCl and will be transported to the endoscopy suite. In the endoscopy suite, the FMT product will be packaged into 6 x 50 ml syringes for patient delivery by colonoscopy.
  Arms: Autologous FMT

SUMMARY:
Every human harbors complex microbial communities (collectively, the human 'microbiome') that cover the skin and the body's mucosal surfaces. There is mounting evidence of an interaction between the intestinal microbiota, the gut, and the central nervous system (CNS) in what is recognized as the microbiome-gut-brain axis. Based on this compelling body of evidence, there is growing enthusiasm for work that is focused on translating this emerging association into novel therapies for psychiatric illness.

Fecal microbiota transplantation(FMT) is a technique in which gut bacteria are transferred from a healthy screened donor to a patient, with the goal to introduce or restore a stable microbial community in the gut.There are no clinical trials examining the impact of FMT on Bipolar Disorder (BD). However, there is biological rationale to support this type of treatment, given the known inflammatory underpinnings of this illness.

The objective of this study is to assess the effectiveness of this very novel therapy targeting the gut-brain axis, FMT, to treat bipolar depression.

Study Hypotheses:

Main hypothesis: FMT from healthy donors to patients with BD depression will improve depression symptoms as an adjunct to approved medication.

Secondary hypotheses:

1. FMT will also reduce anxiety and global function
2. FMT is safe and will be well tolerated by the patients
3. Improvements in clinical parameters will be associated with specific changes in the intestinal microbiome and/or metabolites in stool and serum

DETAILED DESCRIPTION:
The primary goals of this proof of concept study are to determine the effectiveness, safety and tolerability of FMT in adults with BD depression.

Objective 1: To evaluate the effectiveness of the combination of a currently accepted approved therapy for BD depression + FMT in individuals with BD depression. This will be assessed through a change in the Montgomery-Ãsberg Depression Rating Scale (MADRS) total score from baseline (pre-intervention) to the final visit (week 24). The investigators will also assess the proportion of patients withdrawing from study due to inadequate control of depressive symptoms.

Secondary objective 2: To evaluate the effectiveness of FMT on anxiety symptoms and global function/overall improvement in participants with BD depression. Secondary objective 3: To determine the safety and tolerability of FMT in individuals with BD depression. Safety will be evaluated by solicited and unsolicited adverse events, including serious adverse events, throughout the study period. Tolerability will be assessed using the Toronto Side Effect Scale (TSES). This is a 32-item instrument that is designed to establish incidence, frequency, and severity of CNS, gastrointestinal, and sexual side effects.

Secondary objective 4: To assess the effect of FMT on microbiome profile (community structure and functional metagenome) and fecal metabolome. Changes in fecal microbiome profile and fecal metabolome from baseline to the final visit will be assessed using next generation sequencing and nuclear magnetic resonance (NMR) spectrometry, respectively. Changes in mood rating scales will be correlated with a specific microbiome and metabolome signature. Intestinal microbiome and metabolome of healthy donors will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years of age
2. Outpatient status
3. Have a diagnosis of bipolar disorder (BD) (type I or II) according to the Mini International Neuropsychiatric Interview (MINI)
4. Have been on a stable first line treatment for BD depression at an adequate dose for at least 8 weeks prior to study entry
5. Suffer from a current depressive episode (Montgomery-Åsberg Depression Rating Scale (MADRS) score at screening and baseline of ≥ 12)

Exclusion Criteria:

1. DSM-IV criteria for substance abuse within the last 6 months or lifetime dependency
2. Active eating disorders
3. Schizophrenia or schizoaffective disorder
4. Current psychotic symptoms
5. A Young Mania Rating Scale (YMRS) score of ≥12 at screening
6. Active suicidality
7. Regular intake of non-steroidal anti-inflammatory drugs or iron supplements in the 3 months prior to study entry
8. Use of prebiotics or probiotics for medical purposes, use of antibiotics or any experimental drug in the 3 months prior to study entry
9. Chronic gastrointestinal diseases
10. Conditions causing immunosuppression
11. A significant bleeding disorder
12. Any contraindication to colonoscopy
13. Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the MADRS total score from baseline (pre-intervention) to the final visit (week 24). | Every 2 weeks for 24 weeks
  The MADRS score will be used to assess the effectiveness of the combination of a currently accepted approved therapy plus FMT on depression symptoms. The MADRS score will also help assess the percentage of patients who show inadequate control of depressive symptoms

SECONDARY OUTCOMES:
Changes in the the Clinical Global Impression (CGI) scale | Every 2 weeks for 24 weeks
  The effectiveness of Approved treatment + FMT in controlling anxiety symptoms and global function/Overall improvement will be assessed through the CGI
Changes in the the World Health Organization Quality of life (WHOQOL-BREF) rating | Every 2 weeks for 24 weeks
  The effectiveness of Approved treatment + FMT in improving the quality of life of bipolar depression patients will be assessed through the World Health Organization Quality of life (WHOQOL-BREF) questionnaire.
Side effects as reported on the Toronto Side Effect Scale (TSES) | Every 2 weeks for 24 weeks
  The tolerability of FMT will be assessed using the Toronto Side effects Scale (TSES)
Changes in fecal microbiome profile | stool sample collected at Baseline (Visit 2), week 12 and at week 24
  Stool samples will be collected and analysed using next generation sequencing to examine changes in Changes in fecal microbiome profile
Changes in fecal Metabolome | stool sample collected at Baseline (Visit 2), week 12 and at week 24
  Stool samples will be collected and analysed using nuclear magnetic resonance (NMR) spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Taylor, MD, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's college Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
both the descriptive and analyzed data, including individual patient data, will be submitted to the National Database for Clinical Trials related to Mental Illness (NDCT), which is part of the National Institute of Mental Health Data Archive (NDA). The data are de-identified and will be made available to qualified researchers, who have to request access to the dataset.
Supporting Information: CSR
Time Frame: Data will be uploaded every 6 months through the study and released Within 4 months
Access Criteria: Researchers approved for access to NDCT have the ability to download shared data from all clinical trials available in the repository
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Brietzke E, Stertz L, Fernandes BS, Kauer-Sant'anna M, Mascarenhas M, Escosteguy Vargas A, Chies JA, Kapczinski F. Comparison of cytokine levels in depressed, manic and euthymic patients with bipolar disorder. J Affect Disord. 2009 Aug;116(3):214-7. doi: 10.1016/j.jad.2008.12.001. Epub 2009 Feb 28. PMID 19251324
- [Background] Guloksuz S, Cetin EA, Cetin T, Deniz G, Oral ET, Nutt DJ. Cytokine levels in euthymic bipolar patients. J Affect Disord. 2010 Nov;126(3):458-62. doi: 10.1016/j.jad.2010.04.027. PMID 20537397
- [Background] Jiang H, Ling Z, Zhang Y, Mao H, Ma Z, Yin Y, Wang W, Tang W, Tan Z, Shi J, Li L, Ruan B. Altered fecal microbiota composition in patients with major depressive disorder. Brain Behav Immun. 2015 Aug;48:186-94. doi: 10.1016/j.bbi.2015.03.016. Epub 2015 Apr 13. PMID 25882912
- [Background] Naseribafrouei A, Hestad K, Avershina E, Sekelja M, Linlokken A, Wilson R, Rudi K. Correlation between the human fecal microbiota and depression. Neurogastroenterol Motil. 2014 Aug;26(8):1155-62. doi: 10.1111/nmo.12378. Epub 2014 Jun 1. PMID 24888394
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Diaz Heijtz R, Wang S, Anuar F, Qian Y, Bjorkholm B, Samuelsson A, Hibberd ML, Forssberg H, Pettersson S. Normal gut microbiota modulates brain development and behavior. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3047-52. doi: 10.1073/pnas.1010529108. Epub 2011 Jan 31. PMID 21282636
- [Background] Fremont M, Coomans D, Massart S, De Meirleir K. High-throughput 16S rRNA gene sequencing reveals alterations of intestinal microbiota in myalgic encephalomyelitis/chronic fatigue syndrome patients. Anaerobe. 2013 Aug;22:50-6. doi: 10.1016/j.anaerobe.2013.06.002. Epub 2013 Jun 19. PMID 23791918
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Xu MQ, Cao HL, Wang WQ, Wang S, Cao XC, Yan F, Wang BM. Fecal microbiota transplantation broadening its application beyond intestinal disorders. World J Gastroenterol. 2015 Jan 7;21(1):102-11. doi: 10.3748/wjg.v21.i1.102. PMID 25574083
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Zoller V, Laguna AL, Prazeres Da Costa O, Buch T, Goke B, Storr M. [Fecal microbiota transfer (FMT) in a patient with refractory irritable bowel syndrome]. Dtsch Med Wochenschr. 2015 Aug;140(16):1232-6. doi: 10.1055/s-0041-103798. Epub 2015 Aug 11. German. PMID 26261935
- [Background] Colman RJ, Rubin DT. Fecal microbiota transplantation as therapy for inflammatory bowel disease: a systematic review and meta-analysis. J Crohns Colitis. 2014 Dec;8(12):1569-81. doi: 10.1016/j.crohns.2014.08.006. Epub 2014 Sep 13. PMID 25223604
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] EISEMAN B, SILEN W, BASCOM GS, KAUVAR AJ. Fecal enema as an adjunct in the treatment of pseudomembranous enterocolitis. Surgery. 1958 Nov;44(5):854-9. No abstract available. PMID 13592638
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Dickerson FB, Stallings C, Origoni A, Katsafanas E, Savage CL, Schweinfurth LA, Goga J, Khushalani S, Yolken RH. Effect of probiotic supplementation on schizophrenia symptoms and association with gastrointestinal functioning: a randomized, placebo-controlled trial. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01579. doi: 10.4088/PCC.13m01579. Epub 2014 Feb 13. PMID 24940526
- [Background] Rao AV, Bested AC, Beaulne TM, Katzman MA, Iorio C, Berardi JM, Logan AC. A randomized, double-blind, placebo-controlled pilot study of a probiotic in emotional symptoms of chronic fatigue syndrome. Gut Pathog. 2009 Mar 19;1(1):6. doi: 10.1186/1757-4749-1-6. PMID 19338686
- [Background] Logan AC, Katzman M. Major depressive disorder: probiotics may be an adjuvant therapy. Med Hypotheses. 2005;64(3):533-8. doi: 10.1016/j.mehy.2004.08.019. PMID 15617861
- [Background] Girard SA, Bah TM, Kaloustian S, Lada-Moldovan L, Rondeau I, Tompkins TA, Godbout R, Rousseau G. Lactobacillus helveticus and Bifidobacterium longum taken in combination reduce the apoptosis propensity in the limbic system after myocardial infarction in a rat model. Br J Nutr. 2009 Nov;102(10):1420-5. doi: 10.1017/S0007114509990766. Epub 2009 Jun 29. PMID 19563693
- [Background] Sullivan A, Nord CE. Probiotics and gastrointestinal diseases. J Intern Med. 2005 Jan;257(1):78-92. doi: 10.1111/j.1365-2796.2004.01410.x. PMID 15606379
- [Background] Gareau MG, Jury J, MacQueen G, Sherman PM, Perdue MH. Probiotic treatment of rat pups normalises corticosterone release and ameliorates colonic dysfunction induced by maternal separation. Gut. 2007 Nov;56(11):1522-8. doi: 10.1136/gut.2006.117176. Epub 2007 Mar 5. PMID 17339238
- [Background] Eutamene H, Bueno L. Role of probiotics in correcting abnormalities of colonic flora induced by stress. Gut. 2007 Nov;56(11):1495-7. doi: 10.1136/gut.2007.124040. PMID 17938427
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Camilleri M. Probiotics and irritable bowel syndrome: rationale, putative mechanisms, and evidence of clinical efficacy. J Clin Gastroenterol. 2006 Mar;40(3):264-9. doi: 10.1097/00004836-200603000-00020. PMID 16633134
- [Background] Luna RA, Foster JA. Gut brain axis: diet microbiota interactions and implications for modulation of anxiety and depression. Curr Opin Biotechnol. 2015 Apr;32:35-41. doi: 10.1016/j.copbio.2014.10.007. Epub 2014 Nov 21. PMID 25448230
- [Background] Maes M, Kubera M, Leunis JC, Berk M. Increased IgA and IgM responses against gut commensals in chronic depression: further evidence for increased bacterial translocation or leaky gut. J Affect Disord. 2012 Dec 1;141(1):55-62. doi: 10.1016/j.jad.2012.02.023. Epub 2012 Mar 11. PMID 22410503
- [Background] Maes M, Kubera M, Leunis JC. The gut-brain barrier in major depression: intestinal mucosal dysfunction with an increased translocation of LPS from gram negative enterobacteria (leaky gut) plays a role in the inflammatory pathophysiology of depression. Neuro Endocrinol Lett. 2008 Feb;29(1):117-24. PMID 18283240
- [Background] Braniste V, Al-Asmakh M, Kowal C, Anuar F, Abbaspour A, Toth M, Korecka A, Bakocevic N, Ng LG, Kundu P, Gulyas B, Halldin C, Hultenby K, Nilsson H, Hebert H, Volpe BT, Diamond B, Pettersson S. The gut microbiota influences blood-brain barrier permeability in mice. Sci Transl Med. 2014 Nov 19;6(263):263ra158. doi: 10.1126/scitranslmed.3009759. PMID 25411471
- [Background] Collins SM, Surette M, Bercik P. The interplay between the intestinal microbiota and the brain. Nat Rev Microbiol. 2012 Nov;10(11):735-42. doi: 10.1038/nrmicro2876. Epub 2012 Sep 24. PMID 23000955
- [Background] Wang Y, Kasper LH. The role of microbiome in central nervous system disorders. Brain Behav Immun. 2014 May;38:1-12. doi: 10.1016/j.bbi.2013.12.015. Epub 2013 Dec 25. PMID 24370461
- [Background] Petra AI, Panagiotidou S, Hatziagelaki E, Stewart JM, Conti P, Theoharides TC. Gut-Microbiota-Brain Axis and Its Effect on Neuropsychiatric Disorders With Suspected Immune Dysregulation. Clin Ther. 2015 May 1;37(5):984-95. doi: 10.1016/j.clinthera.2015.04.002. PMID 26046241
- [Background] Bangsgaard Bendtsen KM, Krych L, Sorensen DB, Pang W, Nielsen DS, Josefsen K, Hansen LH, Sorensen SJ, Hansen AK. Gut microbiota composition is correlated to grid floor induced stress and behavior in the BALB/c mouse. PLoS One. 2012;7(10):e46231. doi: 10.1371/journal.pone.0046231. Epub 2012 Oct 2. PMID 23056268
- [Background] Judd LL, Akiskal HS, Schettler PJ, Endicott J, Maser J, Solomon DA, Leon AC, Rice JA, Keller MB. The long-term natural history of the weekly symptomatic status of bipolar I disorder. Arch Gen Psychiatry. 2002 Jun;59(6):530-7. doi: 10.1001/archpsyc.59.6.530. PMID 12044195
- [Background] Cryan JF, O'Mahony SM. The microbiome-gut-brain axis: from bowel to behavior. Neurogastroenterol Motil. 2011 Mar;23(3):187-92. doi: 10.1111/j.1365-2982.2010.01664.x. PMID 21303428
- [Background] Forsythe P, Sudo N, Dinan T, Taylor VH, Bienenstock J. Mood and gut feelings. Brain Behav Immun. 2010 Jan;24(1):9-16. doi: 10.1016/j.bbi.2009.05.058. Epub 2009 May 28. PMID 19481599
- [Background] Rhee SH, Pothoulakis C, Mayer EA. Principles and clinical implications of the brain-gut-enteric microbiota axis. Nat Rev Gastroenterol Hepatol. 2009 May;6(5):306-14. doi: 10.1038/nrgastro.2009.35. PMID 19404271
- [Background] Sudo N, Chida Y, Aiba Y, Sonoda J, Oyama N, Yu XN, Kubo C, Koga Y. Postnatal microbial colonization programs the hypothalamic-pituitary-adrenal system for stress response in mice. J Physiol. 2004 Jul 1;558(Pt 1):263-75. doi: 10.1113/jphysiol.2004.063388. Epub 2004 May 7. PMID 15133062
- [Background] Goehler LE, Gaykema RP, Opitz N, Reddaway R, Badr N, Lyte M. Activation in vagal afferents and central autonomic pathways: early responses to intestinal infection with Campylobacter jejuni. Brain Behav Immun. 2005 Jul;19(4):334-44. doi: 10.1016/j.bbi.2004.09.002. PMID 15944073
- [Background] Lyte M, Li W, Opitz N, Gaykema RP, Goehler LE. Induction of anxiety-like behavior in mice during the initial stages of infection with the agent of murine colonic hyperplasia Citrobacter rodentium. Physiol Behav. 2006 Oct 30;89(3):350-7. doi: 10.1016/j.physbeh.2006.06.019. Epub 2006 Aug 2. PMID 16887154
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Kunz M, Cereser KM, Goi PD, Fries GR, Teixeira AL, Fernandes BS, Belmonte-de-Abreu PS, Kauer-Sant'Anna M, Kapczinski F, Gama CS. Serum levels of IL-6, IL-10 and TNF-alpha in patients with bipolar disorder and schizophrenia: differences in pro- and anti-inflammatory balance. Braz J Psychiatry. 2011 Sep;33(3):268-74. doi: 10.1590/s1516-44462011000300010. PMID 21971780
- [Background] Kauer-Sant'Anna M, Kapczinski F, Andreazza AC, Bond DJ, Lam RW, Young LT, Yatham LN. Brain-derived neurotrophic factor and inflammatory markers in patients with early- vs. late-stage bipolar disorder. Int J Neuropsychopharmacol. 2009 May;12(4):447-58. doi: 10.1017/S1461145708009310. Epub 2008 Sep 4. PMID 18771602
- [Background] Desbonnet L, Garrett L, Clarke G, Kiely B, Cryan JF, Dinan TG. Effects of the probiotic Bifidobacterium infantis in the maternal separation model of depression. Neuroscience. 2010 Nov 10;170(4):1179-88. doi: 10.1016/j.neuroscience.2010.08.005. Epub 2010 Aug 6. PMID 20696216
- [Background] Padmos RC, Van Baal GC, Vonk R, Wijkhuijs AJ, Kahn RS, Nolen WA, Drexhage HA. Genetic and environmental influences on pro-inflammatory monocytes in bipolar disorder: a twin study. Arch Gen Psychiatry. 2009 Sep;66(9):957-65. doi: 10.1001/archgenpsychiatry.2009.116. PMID 19736352
- [Background] Baldessarini RJ, Tondo L. Suicide risk and treatments for patients with bipolar disorder. JAMA. 2003 Sep 17;290(11):1517-9. doi: 10.1001/jama.290.11.1517. No abstract available. PMID 13129995
- [Background] Colom F, Vieta E, Martinez-Aran A, Reinares M, Benabarre A, Gasto C. Clinical factors associated with treatment noncompliance in euthymic bipolar patients. J Clin Psychiatry. 2000 Aug;61(8):549-55. doi: 10.4088/jcp.v61n0802. PMID 10982196
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Tang MS, Poles J, Leung JM, Wolff MJ, Davenport M, Lee SC, Lim YA, Chua KH, Loke P, Cho I. Inferred metagenomic comparison of mucosal and fecal microbiota from individuals undergoing routine screening colonoscopy reveals similar differences observed during active inflammation. Gut Microbes. 2015;6(1):48-56. doi: 10.1080/19490976.2014.1000080. Epub 2015 Jan 20. PMID 25559083
- [Background] Parthasarathy G, Chen J, Chen X, Chia N, O'Connor HM, Wolf PG, Gaskins HR, Bharucha AE. Relationship Between Microbiota of the Colonic Mucosa vs Feces and Symptoms, Colonic Transit, and Methane Production in Female Patients With Chronic Constipation. Gastroenterology. 2016 Feb;150(2):367-79.e1. doi: 10.1053/j.gastro.2015.10.005. Epub 2015 Oct 13. PMID 26460205
- [Background] Bajaj JS, Betrapally NS, Hylemon PB, Heuman DM, Daita K, White MB, Unser A, Thacker LR, Sanyal AJ, Kang DJ, Sikaroodi M, Gillevet PM. Salivary microbiota reflects changes in gut microbiota in cirrhosis with hepatic encephalopathy. Hepatology. 2015 Oct;62(4):1260-71. doi: 10.1002/hep.27819. Epub 2015 May 6. PMID 25820757
- [Background] Maynard CL, Elson CO, Hatton RD, Weaver CT. Reciprocal interactions of the intestinal microbiota and immune system. Nature. 2012 Sep 13;489(7415):231-41. doi: 10.1038/nature11551. PMID 22972296
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Vanderkooy JD, Kennedy SH, Bagby RM. Antidepressant side effects in depression patients treated in a naturalistic setting: a study of bupropion, moclobemide, paroxetine, sertraline, and venlafaxine. Can J Psychiatry. 2002 Mar;47(2):174-80. doi: 10.1177/070674370204700208. PMID 11926080
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Drago L, Toscano M, De Grandi R, Casini V, Pace F. Persisting changes of intestinal microbiota after bowel lavage and colonoscopy. Eur J Gastroenterol Hepatol. 2016 May;28(5):532-7. doi: 10.1097/MEG.0000000000000581. PMID 27015015
- [Background] Jalanka J, Salonen A, Salojarvi J, Ritari J, Immonen O, Marciani L, Gowland P, Hoad C, Garsed K, Lam C, Palva A, Spiller RC, de Vos WM. Effects of bowel cleansing on the intestinal microbiota. Gut. 2015 Oct;64(10):1562-8. doi: 10.1136/gutjnl-2014-307240. Epub 2014 Dec 19. PMID 25527456
- [Background] Rossen NG, MacDonald JK, de Vries EM, D'Haens GR, de Vos WM, Zoetendal EG, Ponsioen CY. Fecal microbiota transplantation as novel therapy in gastroenterology: A systematic review. World J Gastroenterol. 2015 May 7;21(17):5359-71. doi: 10.3748/wjg.v21.i17.5359. PMID 25954111
- [Background] Hamilton MJ, Weingarden AR, Unno T, Khoruts A, Sadowsky MJ. High-throughput DNA sequence analysis reveals stable engraftment of gut microbiota following transplantation of previously frozen fecal bacteria. Gut Microbes. 2013 Mar-Apr;4(2):125-35. doi: 10.4161/gmic.23571. Epub 2013 Jan 18. PMID 23333862
- [Derived] Cooke NCA, Bala A, Allard JP, Hota S, Poutanen S, Taylor VH. The safety and efficacy of fecal microbiota transplantation in a population with bipolar disorder during depressive episodes: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Jul 14;7(1):142. doi: 10.1186/s40814-021-00882-4. PMID 34261526
- See also: Microbiota Therapeutics Outcomes Program (MTOP) — https://mtop.ca/funded-projects/